CLINICAL TRIAL: NCT00764959
Title: Post-Market Study of the Linear™ Hip System
Brief Title: Retrospective Study of the Linear™ Hip
Status: Terminated | Type: Observational
Why Stopped: Enrollment and data collection insufficient to continue study.
Sponsor: Encore Medical, L.P. (Industry)
Responsible Party: Jane M. Jacob Ph.D., DJO Surgical
Other Study IDs: PS - 800
Record Dates: First submitted 2008-09-30; First posted 2008-10-02 (Estimated); Last update posted 2011-02-09 (Estimated); Status verified 2011-02

CONDITIONS: Osteoarthritis; Rheumatoid Arthritis; Femoral Fracture; Correction of a Functional Deformity; Avascular Necrosis
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid; Femoral Fractures; Osteonecrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Linear Hip: Encore Linear Hip System
  Interventions: Device: Encore Linear™ Hip System

INTERVENTIONS:
Device: Encore Linear™ Hip System — Subjects with degenerative joint disease (DJD), osteoarthritis or rheumatoid arthritis, have received the hip system and are willing to participate in the study.

SUMMARY:
The purpose of this study is to evaluate the use and efficacy of the Encore Linear™ Hip System in a group of 200 patients for whom data has already been collected.

ELIGIBILITY:
Inclusion Criteria:

* Have hip joint disease related to one or more of the following

  * osteoarthritis
  * rheumatoid arthritis
  * femoral fracture
  * correction of a functional deformity
  * avascular necrosis of the natural femoral head
* Skeletal maturity
* Patient is likely to be available for evaluation for the duration of the study
* Able and willing to sign the informed consent and follow study procedures
* Patient is not pregnant
* No infection present
* No known materials sensitivity
* Patient is over 18 years of age

Exclusion Criteria:

* Skeletal immaturity
* Infection or sepsis
* Insufficient bone quality that may affect the stability of the implant
* Muscular, neurologic or vascular deficiencies which compromise the affected extremity
* Alcoholism or other addictions
* Prisoners
* High levels of physical activity
* Patient is pregnant
* Loss of ligamentous structures
* Materials sensitivity
* Patient is under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals who meet the indications for use of the Linear Hip device AND who meet the inclusion/exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2007-10; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
The use and efficacy of the Encore Linear™ Hip System | 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Omar Hussamy, M.D., Principal Investigator — Hussamy Orthopedics
Locations (1):
- Hussamy Orthopedics, Vero Beach, Florida, United States

REFERENCES:
- See also: Sponsor Company home page — http://www.djosurgical.com